CLINICAL TRIAL: NCT01063153
Title: Diagnostic Utility of ADHD by Brain Activity Flow Patterns Analysis Using Evoked Response Potentials
Brief Title: Diagnostic Utility of Attention Deficit Hyperactivity Disorder (ADHD) by Brain Activity Flow Patterns Analysis Using Evoked Response Potentials
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ElMindA Ltd (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-P-000174
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Adults; Electroencephalography (EEG); Concerta
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concerta (Experimental): Open-Label Concerta (Osmotic Release Methylphenidate)
  Interventions: Drug: Osmotic Release Methylphenidate
- Control group (No Intervention): Healthy subjects without ADHD will be assessed using EEG.

INTERVENTIONS:
Drug: Osmotic Release Methylphenidate — During a 6 week treatment period, adult subjects with ADHD are prescribed, in an open label fashion, once daily doses of osmotic release methylphenidate to a maximum daily dose of 144 mg. Efficacy and tolerability assessments are completed, in addition to EEG and cognitive testing. Healthy adults without ADHD will not receive medication.
  Other Names: Concerta
  Arms: Concerta

SUMMARY:
The purpose of this research study is to study a device called an electroencephalograph (EEG) in the diagnosis of treatment of attention deficit hyperactivity disorder (ADHD) in adults. People with ADHD have symptoms such as difficulty sustaining attention, organizing, and managing impulsivity. They can have trouble in school, at work, and at home. Subjects with ADHD who participate in this study will be given a once daily stimulant medication called osmotic release methylphenidate (Concerta) for 6 weeks, and have EEG testing done before and after the treatment period. Subjects will perform a computer based cognitive task during EEG testing. The U.S. Food and Drug Administration has approved osmotic release methylphenidate (Concerta) for the treatment of ADHD in adults and children. Similar procedures, without medication, will be performed with a sample of healthy adults without ADHD.

ELIGIBILITY:
ADHD Subjects

Inclusion Criteria:

* Male and female outpatients, aged 18-55 years
* Subjects meeting full criteria for the diagnosis of DSM-IV (Diagnostic and Statistical Manual, Version 4) Attention Deficit Hyperactivity Disorder (ADHD)
* Absence of pharmacological treatment for ADHD for at least one week.
* Right handedness

Exclusion Criteria:

* Any other current psychiatric or medical condition determined to be clinically significant.
* Current use of psychotropics or any medication with clinically significant CNS (Central Nervous System) effects.
* Mental retardation (IQ < 80).
* Significant sensory deficits such as deafness or blindness.
* Individuals with a history of substance dependence or abuse within the past 6 months.
* Pregnant or nursing females.
* Subjects with pre-existing structural cardiac abnormalities.
* Clinically significant abnormal laboratory values, electrocardiogram or blood pressure reading

Healthy Control Subjects

Inclusion Criteria:

* Males and females, aged 18-55 years
* Subjects who do not meet full criteria for the diagnosis of DSM-IV Attention Deficit Hyperactivity Disorder (ADHD), as determined by clinical evaluation and/or ADHD module of structured diagnostic interview, completed by the study clinician.
* Right handedness

Exclusion Criteria:

* Any current psychiatric or medical condition determined to be clinically significant.
* Current use of psychotropics or any medication with clinically significant CNS effects.
* Mental retardation (IQ < 80).
* Significant sensory deficits such as deafness or blindness.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Controls without ADHD were assessed using EEG
- ADHD: Subjects with ADHD were assessed with EEG before and after treatment with Concerta
Period: Overall Study
Arm/Group | Control | ADHD
Started | 33 | 38
Completed | 31 | 26
Not Completed | 2 | 12
Not completed — Found Ineligible During Screening | 2 | 0
Not completed — Lost to Follow-up | 0 | 7
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Control: Subjects without ADHD
- ADHD: Subjects with ADHD
- Total: Total of all reporting groups
Arm/Group | Control | ADHD | Total
Number analyzed (Participants) | 33 | 38 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 38 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (11.0) | 35.5 (10.5) | 34.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 17 | 24 | 41
Region of Enrollment [Number; unit: participants]
  United States | 33 | 38 | 71

OUTCOME MEASURES:

1. Primary Outcome: Adult ADHD Investigator Symptom Rating Scale (AISRS)
Description: An 18-item scale rating a subject's level of impairment from 0 (none) to 3 (severe) for each symptom of DSM-IV ADHD, with a maximum possible score of 54. The measure was collected at Baseline and 6 weeks, and a total score was calculated to gauge treatment response of ADHD subjects to open-label Concerta.
Time Frame: Baseline and 6 weeks
Population: Subjects in the ADHD group who completed all 6 weeks of the trial were included in data analysis. Subjects who completed at least 3 weeks of treatment were also included regardless of the reason for withdrawal, and final-visit AISRS scores were used in ITT (intent-to-treat) analysis via last observation carried forward [LOCF] imputation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ADHD: Subjects with ADHD were assessed before and after treatment.
- Controls: Controls without ADHD were assessed with a one-time EEG, only.
Arm/Group | ADHD | Controls
Number analyzed (Participants) | 28 | 0
units on a scale
  Baseline | 37.0 (8.7) |
  6 weeks | 15.0 (9.4) |

2. Primary Outcome: Percent Errors in Visual Go/NoGo Task
Description: The Go/NoGo visual task was completed by subjects with ADHD as well as healthy controls. The Go/NoGo task is used to assess inhibitory control, and targets response inhibition, executive functions, and sustained attention. The 'Go' stimulus occupies 80% of the trials, and requires the subject to perform a motor response each time it appears on the screen. A rare 'No Go' stimulus (occupies 20% of all trials) requires the subject to refrain from responding. The percentage of errors were measured for each group.
Time Frame: Single Point (Baseline)
Population: Only subjects that met the a priori pre-defined EEG signal quality criteria were included.
Measure: Number; unit: percentage of errors
Groups:
- ADHD and Visual NoGo Task: Participants with a DSM-IV diagnosis of ADHD completed the NoGo Visual Task, in which they had to refrain from responding.
- Control Group and Visual NoGo Task: Participants without a DSM-IV diagnosis of ADHD completed the NoGo Visual Task, in which they had to refrain from responding.
- ADHD and Visual Go Task: Participants with a DSM-IV diagnosis of ADHD completed the Go Visual Task, in which they had to perform a motor response to a stimulus.
- Control Group and Visual Go Task: Participants without a DSM-IV diagnosis of ADHD completed the Go Visual Task, in which they had to perform a motor response to a stimulus.
Arm/Group | ADHD and Visual NoGo Task | Control Group and Visual NoGo Task | ADHD and Visual Go Task | Control Group and Visual Go Task
Number analyzed (Participants) | 26 | 27 | 30 | 26
percentage of errors | 19.01 | 13.89 | 2.88 | 1.27

ADVERSE EVENTS:
Groups:
- Control: Subjects without ADHD were assessed using EEG.
- ADHD: Subjects with ADHD were assessed with EEG before and after open-label treatment with Concerta.
Arm/Group | Control | ADHD
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/38
Other Adverse Events (participants affected / at risk) | 0/33 | 22/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=33) | ADHD (N=38)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 9 (20)
Dry Mouth (General disorders) | 0 (0) | 2 (5)
Dulled Affect (Psychiatric disorders) | 0 (0) | 4 (5)
Gastrointestinal Upset (Gastrointestinal disorders) | 0 (0) | 3 (3)
Headache (General disorders) | 0 (0) | 11 (19)
Racing Heart (Cardiac disorders) | 0 (0) | 3 (5)
Increased Energy (General disorders) | 0 (0) | 3 (5)
Irritability (General disorders) | 0 (0) | 3 (7)
Jitteriness (General disorders) | 0 (0) | 4 (7)
Tiredness (General disorders) | 0 (0) | 4 (8)
Tension (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Brain Network Analysis [the primary analysis of EEG data related to BAFPA (Brain Activity Flow Patterns Analysis) and functional connectivity networks] is still in progress by the Sponsor, and there is an agreement between the Sponsor and the Principal Investigator preventing the PI from disclosing EEG results from this trial until the data has been published. We are, however, at liberty to report adverse events from the open-label clinical trial and have done so here.